CLINICAL TRIAL: NCT02165800
Title: Multicenter Study on Outcomes and Protection of Urinary and Sexual Function of Laparoscopic Versus Open PANP-TME for Male Mid-low Rectal Cancer Patients
Brief Title: Multicenter Study on Laparoscopic Versus Open PANP-TME for Male Mid-low Rectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Nanfang Hospital, Southern Medical University (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Chief of surgery, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUSTOMER-001
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Rectum Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- O-PANP-TME (Active Comparator): Open pelvic autonomic nerve preservation total mesorectum excision for male mid-low rectal cancer patients
  Interventions: Procedure: O-PANP-TME
- L-PANP-TME (Experimental): Laparoscopy-assisted pelvic autonomic nerve preservation total mesorectum excision for male mid-low rectal cancer patients
  Interventions: Procedure: L-PANP-TME

INTERVENTIONS:
Procedure: L-PANP-TME
  Arms: L-PANP-TME
Procedure: O-PANP-TME
  Arms: O-PANP-TME

SUMMARY:
TME (Total mesorectum excision) is the golden standard of radical resection for mid-low rectal cancer. However, the damage of pelvic autonomic nerve following with TME principle will lead to high incidence of urinary and sexual function disorder. Open PANP (pelvic autonomic nerve preservation) TME surgery played a role in decreasing incidence of urinary and sexual function disorder. However, 32%-44% patients still suffered from urinary and sexual function disorder when underwent Open PANP TME surgery (O-PANP-TME).

Laparoscopy-assisted TME surgery (L-TME) is applied wildly nowadays. In the early stage of work, we performed laparoscopy-assisted PANP TME surgery (L-PANP-TME) to discuss the protection of urinary and sexual function of male mid-low rectal cancer patients. The results showed that L-PANP-TME significantly decreased incidence of urinary and sexual function disorder. In order to further confirm our early work, we design a multiple-center randomized controlled clinical trial to compare differences in urinary and sexual function protection and long-term outcomes between L-PANP-TME and O-PANP-TME.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 20 to under 60 years
* Primary rectal adenocarcinoma confirmed pathologically by endoscopic biopsy
* Mid-low rectal cancer (distance from anal edge≤12cm); cT1-3, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition
* Expected curative resection through both L-PANP-TME and O-PANP-TME; Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I, II, or III; Written informed consent
* Urinary and sexual function normal preoperatively

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous pelvic surgery
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Contraindication of heart, brain, lung, etc dysfunction
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by rectal cancer
* Rectal cancer invades surrounding tissues
* Existence of genuine incontinence or severe stress incontinence preoperatively

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 667 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
Urinary function | 30 days
  Urodynamic study and IPSS (International prostate symptom score) are used to assess urinary function
Sexual function | 30 days
  IIEF-5 (International questionnaire of erectile function-5) and Ejaculation function classification are used to assess sexual function
5-year disease free survival rate | 60 months
Urinary function | 36 months
  Urodynamic study and IPSS (International prostate symptom score) are used to assess urinary function
Sexual function | 36 months
  IIEF-5 (International questionnaire of erectile function-5) and Ejaculation function classification are used to assess sexual function

SECONDARY OUTCOMES:
Morbidity | 30 days
3-year overall survival rate | 36 months
Mortality | 30 days
Morbidity | 36 months
Mortality | 36 months
5-year overall survival rate | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China